CLINICAL TRIAL: NCT06296537
Title: Comparison of the Effectiveness of Balance Training and Dynamic Neuromuscular Stabilization Training in Amateur Athletes with Chronic Ankle Instability
Brief Title: Effectiveness of Balance Training and Dynamic Neuromuscular Stabilization Training in Amateur Athletes with Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Sevval Yesilkır, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-1434
Record Dates: First submitted 2024-02-29; First posted 2024-03-06 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Ankle Inversion Sprain; Chronic Instability of Joint; Chronic Pain; Athlete Foot
Keywords: Chronic Ankle Instability; Dynamic Neuromuscular Stabilization Training; Balance Training; Amateur Athletes; Stabilization
MeSH Terms: conditions — Chronic Pain; Tinea Pedis

STUDY DESIGN:
Intervention Model Description: It is designed as a prospective, randomized, controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dynamic Neuromuscular Stabilization Training Group (Experimental): A dynamic neuromuscular stabilization training program consisting of a series of special exercises based on the developmental kinesiology steps of a healthy baby will be prepared and applied for athletes in the DNS group. As the sessions progress, elastic bands will be used to create resistance in the exercises as the participants gain stabilization. All exercises will start with 1 set of 3 repetitions and increase to 1 set of 20 repetitions. All exercises will be performed barefoot.
  Interventions: Procedure: Dynamic Neuromuscular Stabilization Training (DNS)
- Balance Training Group (Experimental): An intervention program will be prepared for balance training group in which balance training is added to an effective postural stability program. As the sessions progress, hand and ankle sandbags will be used together with the exercises. All exercises will start with 1 set of 10 repetitions and increase to 3 sets of 15 repetitions. Exercises will be performed barefoot.
  Interventions: Procedure: Balance Training
- Conventional Training Group (Active Comparator): A program including stretching, joint range of motion, strengthening and postural control exercises will be prepared for athletes in the conventional group. As the sessions progress, hand and ankle sandbags will be used together with the exercises. All exercises will start with 1 set of 10 repetitions and increase to 3 sets of 15 repetitions. Exercises will be performed barefoot.
  Interventions: Procedure: Conventional Training

INTERVENTIONS:
Procedure: Dynamic Neuromuscular Stabilization Training (DNS) — Dynamic neuromuscular stabilization training has been developed, which optimizes the movement system based on the scientific principles of developmental kinesiology. DNS training aims to stimulate the natural movement control system in the brain to activate the body's stabilization system. Supine, prone, oblique sitting, tripod, high kneeling, hanging stance-midstance faze, hanging stance- propulsion, bear, squat exercises will be applied.
  Arms: Dynamic Neuromuscular Stabilization Training Group
Procedure: Balance Training — Multi-plane single limb challenges, jumping and landing exercises, proprioceptive exercises, and perturbation exercises
  Arms: Balance Training Group
Procedure: Conventional Training — Education, electrotherapy, soft tissue fascia massage, stretching, range of motion, strengthening and postural control exercises
  Arms: Conventional Training Group

SUMMARY:
The goal of this clinical trial is to determine and compare the effects of balance and dynamic neuromuscular stabilization training on ankle function ability, functional instability severity, physical activity level, muscle strength, proprioception, stabilization, balance, reaction time and performance of amateur athletes with chronic ankle instability. The main questions it aims to answer are:

* Do balance and dynamic neuromuscular stabilization training positively affect functionality, balance, stabilization, proprioception and performance in amateur athletes with chronic ankle sprains?
* Does balance training or dynamic neuromuscular stabilization training have a more positive effect on functionality, balance, stabilization, proprioception and performance in amateur athletes with chronic ankle sprains?

Participants will apply:

* a dynamic neuromuscular stabilization training program consisting of a series of special exercises based on the developmental kinesiology steps of a healthy baby.
* balance training which consist of an effective postural stability program.
* conventional training program which consist of stretching, joint range of motion, strengthening and postural control exercises.

Researchers will compare balance and dynamic neuromuscular stabilization training to see if effectiveness of ankle function ability, functional instability severity, physical activity level, muscle strength, proprioception, stabilization, balance, reaction time and performance.

DETAILED DESCRIPTION:
Chronic ankle instability is a repetitive chronic ankle imbalance that leads to a high rate of ankle sprains. Ankle sprains remain the most common foot-ankle and sports injury for which individuals require medical care, including emergency room visits. It is known that 58.5% of professional basketball and football athletes experience ankle sprains. Approximately three-quarters of patients who sustain an ankle sprain have persistent symptoms 1.5 to 4 years after the injury.

The hallmark symptoms of chronic ankle instability are a history of recurrent sprains and/or repeated episodes of giving-way and/or a feeling of instability. Additionally, many permanent symptoms such as pain, structural changes, and adaptations in the sensorimotor and vestibular systems have also been reported. Both acute trauma and residual neuromuscular adaptations lead to biomechanical changes, resulting in chronic ankle instability. Chronic ankle instability generally occurs as a result of 2 deficiencies: functional instability caused by proprioceptive and neuromuscular deficiencies and mechanical instability caused by changes in joint structure and function.

Lateral ankle sprains and chronic ankle instability cause changes in feedback control, which regulates motor control through reflex loops, and in feedforward control, which plans the movement pattern based on especially past experience. Due to changes in neuromuscular control, kinematic and kinetic adaptations are also common in individuals with chronic ankle instability compared to uninjured individuals, and these adaptations may result in abnormal tension on the talar joint cartilage. Therefore, there is a need to identify therapeutic interventions that can restore appropriate neuromuscular control strategies.

Surgical and conservative treatment methods that assist in ankle-foot deformity recovery, return to social life activities and return to sports can provide even better results with in-depth knowledge of ankle anatomy, biomechanics and pathology. Anatomical repair, tendon augmentation, or both are the basic methods of surgical intervention, and today, arthroscopy treatment is becoming more and more common in the treatment of chronic ankle instability. Conservative treatments include the use of orthoses in the acute period and physical therapy modalities that can be applied in the acute/chronic period . Exercise therapy in physiotherapy is one of the most supported interventions in treating chronic ankle instability and significantly reduces the risk of re-injury. Strength training, balance and dual task training, and isokinetic exercises are effective in ankle instability. It has been reported that 6 weeks of dynamic neuromuscular exercise training leads to improvements in sensorimotor control of the ankle joint in athletes with chronic ankle instability. Moreover, balance training exercises based on multi-station tasks have been observed to significantly improve self-reported sense of instability and dynamic balance in individuals with chronic ankle instability. It has been reported that rehabilitation protocols focusing on balance training effectively improve health-related quality of life in individuals with chronic ankle instability. However, it is recommended that interventions include more open chain joint position sense training, multi-plane single limb challenges, and jumping and landing exercises. In addition, during rehabilitation, the focus should not only be on exercising the muscles in their dynamic anatomical functions, but their stabilizing functions should also be addressed. Therefore, dynamic neuromuscular stabilization (DNS) training has been developed, which optimizes the movement system based on the scientific principles of developmental kinesiology. DNS training aims to stimulate the natural movement control system in the brain to activate the body's stabilization system. In the literature, studies on the effects of DNS training on ankle sensorimotor control and ankle joint position are limited. Our aim in this study is to determine and compare the effects of balance and DNS training on ankle function adequacy, functional instability severity, physical activity level, muscle strength, proprioception, stabilization, balance, reaction time and performance of amateur athletes with chronic ankle instability.

Our hypothesis in this study:

H0: Balance and DNS training does not positively affect functionality, balance, stabilization, proprioception and performance in amateur athletes with chronic ankle sprains.

H1: Balance and DNS training positively affects functionality, balance, stabilization, proprioception and performance in amateur athletes with chronic ankle sprains. The effect of balance training is superior to DNS training.

H2: Balance and DNS training positively affects functionality, balance, stabilization, proprioception and performance in amateur athletes with chronic ankle sprains. The effect of DNS training is superior to balance training.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being a non-smoker
* Being an athlete at amateur level
* Score 25 or less on the Cumberland Ankle Instability Questionnaire
* At least 1 acute ankle inversion sprain resulting in swelling, pain, and dysfunction that occurred at least 12 months before the study
* Feeling of giving way in the ankle at least 2 times in the last 6 months

Exclusion Criteria:

* If the patient has any mental problems
* Neurological diseases
* Cerebellar, vestibular, cochlear and inner ear dysfunction
* Surgeries on musculoskeletal structures, chronic musculoskeletal disorders, severe acute lower extremity injuries or head trauma in the last 6 months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-11 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Star Excursion Balance Test | Beginning of the study, and 6th week and 12th week after beginning the study
  The star excursion balance test is a test used to evaluate dynamic balance and dynamic postural stability. A small number of material installations are required to perform the star balance test. Four strips of athletic tape will each need to be cut to lengths ranging from 182.88 cm to 243.84 cm. Two pieces will be used to form a "+", the other two will be placed on top to form an "x", creating a star shape. All lines will be separated from each other at a 45° angle. The participant will maintain balance on the one foot while using other foot to reach as far as possible in 8 different directions. The participant will reach with his feet in 8 different directions: anterior, anteromedial, medial, posteromedial, posterior, posterolateral, lateral and anterolateral.
Balance Error Scoring System (BESS) | Beginning of the study, and 6th week and 12th week after beginning the study
  BESS is a reliable and inexpensive tool to measure static balance in people with chronic foot instability. BESS consists of 6 tests that include both leg stance, one leg stance and tandem stance conditions, respectively, on both hard and foam surfaces with eyes closed. A stopwatch is used to determine participants' time during 20-second stance tests. The grading method is based on the score of the error table in the six tests. Errors include lifting the hip, walking, opening the eyes, grasping something, falling, leaving the test position after 5 seconds, flexion or abduction of the upper leg more than 30 degrees, and lifting the heel or front of the leg on the surface. If more than one mistake is made at the same time, they are counted as one mistake. The maximum total number of errors for any test is taken to be 10.

SECONDARY OUTCOMES:
Foot and Ankle Ability Measurement (FAAM) | Beginning of the study, and 6th week and 12th week after beginning the study
  The foot and ankle ability measure was designed by R. Martin and colleagues in 2005 to detect changes in ankle function over time. It is a self-report questionnaire consisting of two subscales: activities of daily living (ADL) (FAAM, 21 items) and sports (FAAM-S, 8 items). ADL and Sports subscales are scored separately. The response to each item on the ADL subscale is scored from 4 to 0, with 4 meaning "no difficulty" and 0 meaning "cannot do." If the subject answers all 21 items, the highest potential score is 84. The sport subscale is scored in the same way, with 4 meaning 'no difficulty' and 0 meaning 'can't do'. If the subject answers all 8 items, the highest potential score is 32. The Turkish validity and reliability study of the Foot and Ankle Ability Measurement by Çelik et al. has been accepted.
Cumberland Ankle Instability Questionnaire | Beginning of the study, and 6th week and 12th week after beginning the study
  The CAIT, which includes a 9-item 30-point scale, is an effective tool for assessing the severity of functional instability, monitoring progress, and measuring treatment outcome. Participants with a score of 25 or higher are less likely to have functional instability, while participants with a score of 25 or lower are more likely to have functional instability. The Turkish validity and reliability study of the Cumberland Ankle Instability Questionnaire by Candeniz et al. has been accepted.
International Physical Activity Questionnaire - Short Form | Beginning of the study, and 6th week and 12th week after beginning the study
  The International Physical Activity Questionnaire-Short Form assesses the number of days and time spent on moderate to vigorous physical activity, walking and sitting, performed for at least 10 minutes in the previous 7 days. The survey consists of 7 open-ended questions. The summary score is expressed in physical activity metabolic equivalent task-minutes (MET-min/week) per day or week. The scores are calculated as follows: Walking MET-min/week = 3.3 X walking minutes X number of walking days; moderate MET-min/week = 4.0 X minutes of moderate activity X number of days of moderate activity; vigorous MET-min/week = 8.0 X minutes of vigorous activity X number of days of vigorous activity. The short form is preferred because it is easy to administer and shows similar reliability and validity results compared to the long form. The validity and reliability study of the International Physical Activity Questionnaire- Short Form Turkish by Sağlam et al. has been accepted.
Manual Muscle Strength Test with Hand Dynamometer | Beginning of the study, and 6th week and 12th week after beginning the study
  A hand dynamometer is used to assess isometric muscle strength. Muscle forces are tested in four directions: dorsiflexion, plantar flexion, inversion and eversion. Participants are placed in the subtalar neutral position for all tests. The untested leg is stabilized with straps to stabilize and prevent any accessory movement. The hand dynamometer is calibrated and placed on the upper part of the metatarsal heads depending on the position of the foot. Participants are instructed to pull or push the device as hard as possible in each direction, and the researcher responds to this force with both hands for 3 seconds per trial. Three consecutive trials are performed with a 10-second rest between trials. Maximum force as the participant's highest force is used for analysis. All manual muscle testing movements and positions were consistent with the procedures outlined by Daniels and Worthingham
Single Heel Lift Test | Beginning of the study, and 6th week and 12th week after beginning the study
  The test is a modification of the method described by Lunsford and Perry for assessing static ankle balance. Participants stand away from the researcher. They are asked to simply stand on their affected leg, then plantar flex the ankle and elevate on their toes. The test ends when the heel touches the ground. The time the heel touches the ground is recorded. The single heel lift test is the most reliable test reflecting the lack of inversion strength in chronic foot instability.
Joint Position Sense Test | Beginning of the study, and 6th week and 12th week after beginning the study
  Joint position sense is assessed by passively or actively placing the participant's ankle in three different degrees of inversion. These degrees are increments of 30, 60, and 90 percent of the participant's maximum ankle inversion active range of motion in the position where the ankle is at 42 degrees of plantarflexion. The participant is given three seconds to register the position before the ankle returns to the starting position. In the passive test, the ankle is passively moved into inversion at the same movement speed and the participant is asked to say "stop" when he perceives that the test position has been reached. If the participant feels that they are out of position, the ankle is passively rotated back to correct this. In active testing, the participant performs an active inversion movement aimed at stopping the movement in the test position. The order of the test, three different positions and two different methods, is chosen randomly.
Foot Lift Test | Beginning of the study, and 6th week and 12th week after beginning the study
  The participant performs a single-leg stance on the affected leg with eyes closed. The participant stands upright with his/her hands on the hips, spine erect, and head facing forward. The test is performed for 30 seconds and the number of foot lifts during each trial is recorded. Foot lift is defined as any part of the foot leaving the ground. Touching the ground with the opposite foot is recorded as an error. Participants are instructed not to take their hands off their hips, not to open their eyes, and not to touch their stance limb with the opposite foot; however, these actions are not recorded as errors. A single test trial is allowed for participants to acclimate before the test trials. The test is performed 3 times with a 30-second rest between trials. The trial with the most errors is used for analysis.
Blazepod Reaction Time | Beginning of the study, and 6th week and 12th week after beginning the study
  Blazepod reaction time, a new technology, is related to how quickly athletes react to a visual stimulus. The participant stands in the middle of the square shape placed on the ground. A blazepod is placed in each corner of the square. The distance between each blazepod will be equal to the length of the participant's lower extremity. The aim of this test is to reach as much light as possible with the affected foot for 30 seconds, with a one-legged balance activity. Three trials are performed and the best value obtained is recorded. A one-minute rest interval is given between all trials.
Side Hop Test | Beginning of the study, and 6th week and 12th week after beginning the study
  The side hop test is applied to evaluate the participant's functional performance. The participant performs 10 jumps medially and laterally over a 3 cm line on one foot. Ten jumps are performed as quickly as possible. The time to perform the test is measured using a handheld stopwatch. The test is performed twice on the affected limb, with a 60-second rest between trials. The shortest trial is used for analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Sevval Yeşilkır, Istanbul, Beşiktaş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yesilkir S, Ergezen Sahin G. Dynamic neuromuscular stabilization, balance, and conventional training for chronic ankle instability in amateur athletes: a randomised controlled trial. BMC Sports Sci Med Rehabil. 2025 Oct 1;17(1):286. doi: 10.1186/s13102-025-01319-8. PMID 41035081